CLINICAL TRIAL: NCT05031182
Title: Tolerance of the vNOTES Surgical Technique in Total Hysterectomy for Benign Lesion. Clinical Trial of Non-inferiority Compared to the Laparoscopic Technique.
Acronym: VLAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2021 CURINIER; 2021-A01218-33 (Other: 2021-A01218-33)
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-03

CONDITIONS: Hysterectomy; Laparoscopy; vNOTES
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopy (Placebo Comparator): In this Arm, patient will have the traditional hysterectomy by laparoscopy. This is the type of surgery that we realize everyday.
  Interventions: Procedure: Laparoscopy
- vNOTES (Active Comparator): In this Arm, patient will have the hysterectomy by vNOTES (vaginal natural orifices Transluminal surgery). It's the new type of surgery that we want prove the no-inferiority.
  Interventions: Procedure: vNOTES

INTERVENTIONS:
Procedure: Laparoscopy — The hysterectomy is performed by laparoscopy as described in the EMC.
  Arms: Laparoscopy
Procedure: vNOTES — The hysterectomy is performed by vNOTES as described Dr BAEKELANDT and this team.
  Arms: vNOTES

SUMMARY:
During a first consultation with an indication of total hysterectomy for a benign lesion, we will study the patient's eligibility. After explanations of the study and submission of the forms, the patient will benefit from a second consultation with the investigator to give her consent. The surgeon will randomize the patient using RedCap computer software. The patient will then be referred either to the vNOTES group or to the laparoscopy group. The surgery will be performed by surgeons called "expert" in one of the ways first. For this, it will be necessary to have performed at least 25 hysterectomies by laparoscopy or vNOTES. The surgery will take place using the usual techniques. Per and postoperative complications will be studied and noted up to six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman eligible for total hysterectomy for benign lesions with or without bilateral adnexectomy.
* Able to give informed consent to participate in research.
* Affiliation to a Social Security scheme.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Contraindication to the laparoscopic approach
* Contraindication to first vNOTES, in particular: virginity, history of rectal surgery, rectovaginal endometriosis, high active genital infection
* Indications for another concomitant surgical procedure (other than procedure on the appendix)
* Indication of hysterectomy for malignant lesion.
* Any concomitant pathology deemed incompatible with the study.
* COVID not cured or SARS-COv2 positivity dating less than 3 days before surgery.
* Adult patient protected, under guardianship or curatorship or legal safeguard
* Refusal of participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Complications per or post Operative | one month after surgery
  Appearance of a per or post operative complication: bleeding, digestive or urinary sore or infection

SECONDARY OUTCOMES:
Measure of pain | Until one month
  Quantification of postoperative pain: 6 hours, 24 hours, day 2, 5, 7, 14 and at one month
Duration of operation | one day
  From skin opening to skin or vaginal closure
Assessment of quality of life | Six month
  Respond to SF-36 questionnaire to assess and compare quality of life before and after surgery
Assessment of satisfaction | Six month
  Respond to FSFI questionnaire to assess and compare sexuality before and after surgery
Duration of work stoppage | one month
  Patients will inquire if they needed to prolong the sick leave.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra CURINIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU clermont-ferrand, Clermont-Ferrand
  - CH d'Issoire, Issoire

REFERENCES:
- [Derived] Pickett CM, Seeratan DD, Mol BWJ, Nieboer TE, Johnson N, Bonestroo T, Aarts JW. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2023 Aug 29;8(8):CD003677. doi: 10.1002/14651858.CD003677.pub6. PMID 37642285